CLINICAL TRIAL: NCT06903962
Title: Mind Body Intervention for Chronic Upper Extremity Pain (Repetitive Stress Injury)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000579
Record Dates: First submitted 2025-03-26; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain; Chronic Pain Syndrome; Repetitive Stress Injury
MeSH Terms: conditions — Chronic Pain; Cumulative Trauma Disorders

STUDY DESIGN:
Intervention Model Description: This is a cohort study in which all participants will receive the mind-body intervention. We will not modify participant medication regimens and no pain or other medication prescriptions will be issued by the research team at any time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Mind-body Intervention (Experimental): Mind body techniques for the intervention will be taught in lectures and group discussion sessions
  Interventions: Behavioral: Mind-Body Intervention

INTERVENTIONS:
Behavioral: Mind-Body Intervention — The mind-body intervention will include regular approximate 2 hour educational sessions and didactics learning mind body techniques. The sessions will be twice per week for the first 4 weeks and then subsequently once per week for a total of 13 weeks.

SUMMARY:
The goal of this nonrandomized pilot study is to test a mind-body interventional approach for the treatment of chronic upper extremity pain or repetitive stress injury of the upper extremity (wrist/shoulder/elbow).

1. To determine if a mind-body intervention improves upper extremity functional capacity (ie., Disability of Arm Shoulder Hand - DASH) among people with chronic wrist, elbow, and shoulder pain
2. To determine if a mind-body intervention decreases pain intensity, pain-related anxiety, and overall somatic complaints in our trial participants.
3. To tailor the intervention and the outcomes assessment procedures for conducting a trial in a population with upper extremity pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years of age)
2. A disability score ≥ 40 as per the QuickDASH survey
3. Presence of pain and perceived disability for a minimum of 3 months
4. Willing to engage in a Mind-Body intervention
5. Positive visualization test (onset of pain when patients visualize themselves performing tasks that generally bring on pain)

Exclusion Criteria:

1. Clear organic diagnosis of pain (e.g., cancer, infection, etc…) not inclusive of non-specific findings on imaging studies (e.g., mild arthritis)
2. Age greater than 60 years (due to an increased risk of there being an organic/physical cause for their pain and confounding results)
3. Diagnosis of cognitive impairment or dementia
4. Active addiction disorder, e.g. cocaine or IV heroin use, that would interfere with study participation
5. Major psychiatric comorbidity (e.g., schizophrenia). Anxiety and mild-moderate depression are not considered in this category

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) | Baseline, 4 weeks, 8 weeks, 13 weeks
  The DASH is a commonly used and validated 38 question survey self-report survey assessing the effects of upper extremity disabling conditions on functional activity, pain, sleep, and other parameters

SECONDARY OUTCOMES:
Upper Extremity Function Scale | Baseline, 4 weeks, 8 weeks, 13 weeks
  The Upper Extremity Function Scale is an alternative instrument to the DASH which contains both common and unique evaluation questions.
Brief Pain Inventory Questionnaire (Short Form) | Baseline, 4 weeks, 8 weeks, 13 weeks
  The Brief Pain Inventory questionnaire will be utilized to gauge pain intensity during the duration of the study.
Pain Anxiety Symptom Scale (short form 20) | Baseline, 4 weeks, 8 weeks, 13 weeks
  The short form Pain Anxiety Symptom Scale (PASS-20) is a 20 question survey assessing cognitive, avoidance, fear, and physiological anxiety due to pain.
Somatic Symptom Score (SSS-8) | Baseline, 4 weeks, 8 weeks, 13 weeks
  The 8 question SSS-8 is an abbreviated version of the 15 question Patient Health Questionnaire (PHQ)-15. SSS-8 survey questions pertain to pain, the gastrointestinal system, fatigue, and cardiovascular complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No